CLINICAL TRIAL: NCT06503575
Title: Investigation of Body Schema as Sensorimotor Representation in Adolescent Idiopathic Scoliosis and Comparison With Healthy Individuals-A Case Control Study
Brief Title: Adolescent Idiopathic Scoliosis and Body Schema
Status: Not yet recruiting | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assoc, Prof. Nuray Alaca, Head of department Physiotherapy and Rehabilitation, Acibadem University
Other Study IDs: ATADEK-2024/9/343
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Adolescent Idiopathic Scoliosis; Body Schema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with adolescent idiopathic scoliosis
  Interventions: Other: Assesment
- Healthy control
  Interventions: Other: Assesment

INTERVENTIONS:
Other: Assesment — All assessments will be made

SUMMARY:
Adolescent idiopathic scoliosis is the most common form of scoliosis. Although an increasing number of studies suggest that an abnormal sensory-motor integration critically contributes to the cause of adolescent idiopathic scoliosis , there is uncertainty about the level of the central nervous system explaining this dysfunction. Therefore, the planned master's thesis study aims to compare proprioception, tactile acuity, right-left reasoning ability, motor imagery ability, including the evaluation of body schema, which is a sensorimotor representation in adolescent idiopathic scoliosis patients with healthy individuals. In addition, the relationship of these markers with posture results, body perception and quality of life of individuals with adolescent idiopathic scoliosis will be investigated as a secondary aim.

ELIGIBILITY:
Inclusion Criteria (Adolescent idiopathic scoliosis)

* Diagnosis of Adolescent idiopathic scoliosis
* Age ⩾19 years old
* Curve severity over 10°

Exclusion Criteria (Adolescent idiopathic scoliosis)

* History of spine surgery
* Surgery or trauma
* Secondary scoliosis
* Unable to fill out the questionnaires or attend the physical examination,
* History of musculoskeletal injury in the last six months
* Known systematic and psychological illness
* Use of prescription medication

Inclusion Criteria (adolescent healthy/untreated population)

-Age ⩾ 19 years Matched for age/height/weight (+/-5 years; +/- 10 lbs; +/- 10cm) to a scoliosis participant

Exclusion Criteria (adolescent healthy/untreated population)

* History of spine surgery
* Spine deformity
* Surgery or trauma
* Primer and Secondary scoliosis
* Unable to fill out the questionnaires or attend the physical examination,
* History of musculoskeletal injury in the last six months
* Known systematic and psychological illness
* Use of prescription medication

Ages: 11 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescent idiopathic scoliosis consulting a surgeon and adolescent healthy/untreated population consulting a surgeon
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
The two-point discrimination test | Baseline
  The two-point discrimination test is used to assess if the patient is able to identify two close points on a small area of skin, and how fine the ability to discriminate this are. It is a measure of tactile agnosia, or the inability to recognize these two points despite intact cutaneous sensation and proprioception
Left/right discrimination (Lateralization) | Baseline
  Right-Left Discrimination will be evaluated with Recognise™ applications (Back) developed by the "Neuro Orthopedic Institute".
Kinesthetic and Visual Imagery Questionnaire | Baseline
  Motor imagery ability will be assessed with the Kinesthetic and Visual Imagery Questionnaire (KVIQ). The participant gives a score between 1 and 5 for the image he/she imagines: "1 point: no image, 5 points: as clear as the original." This process is repeated for each task and at the end of the survey, kinesthetic imagery score, visual imagery score and total score are calculated.
Lumbar proprioception test | Baseline
  In both groups, thoracic and lumbar repositioning accuracy will be measured and evaluated using the dual inclinometer system.
Pressure Pain Threshold | Baseline
  A digital pressure algometer will be applied to the web space of the foot opposite the trigger point. Participants are instructed to say "stop" or "pain" so the stimulus can be terminated "when the sensation first transitions from pressure to pain" (pain threshold).

SECONDARY OUTCOMES:
4D DIERS FORMETIC | baseline
  In this study, the newly developed 4D DIERS FORMETIC movable spine and surface topography evaluation device will be used. This device is equipped with a digital network camera that allows measurements at a maximum frequency of up to 50 frames per second. The camera uses CMOS sensors with a resolution of 1280x1024 pixels. Thanks to these sensors and reflective markers, measurements are reconstructed in 3D. Thus, it allows real-time evaluation of posture parameters. Evaluation is done without radiation and without contact.
Body Image Disturbance Questionnaire--Scoliosis Version | Baseline
  It is a seven-item instrument that measures body image disturbance. It assesses (1) concern about body part(s) felt to be unattractive; (2) preoccupation with the concern(s); (3) experiences of emotional distress about appearance; (4) impairment in social, occupational, or other areas of functioning; (5) interference with social life, school, job, or role functioning; (6) avoidance of activities because of appearance; and (7) behavioral avoidance10,26. Using a rating scale from 1 to 5 (with 1 = not at all concerned, and 5 = extremely concerned) to measure each of these items and a mean score for the seven items, the BIDQ allows for continuous, quantitative measurement. Higher scores reflect more severe body image disturbance
Walter Reed Visual Assessment Scale | Baseline
  It is a scale that scores the severity of curvature by focusing on the person's perception of posture. It is divided into 7 parameters including body curvature, rib prominence, lumbar prominence, head-rib-pelvis positional relationship, head-pelvis relationship, shoulder level and scapula rotation. A high score means that the perceived deformity is high.
Scoliosis Research Society 22 | Baseline
  It is a quality of life questionnaire which consists of 22 questions assessing 5 quality of life domains: Function, Pain, Self-Image, Mental health (5 questions), satisfaction (2 questions). Each category is rated on 5. The categories are summed and divided by 5 to have a total score on 5 points. 5 is the best score and 1 the worst

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acibadem University, Istanbul
  - Maslak Acıbadem, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided